CLINICAL TRIAL: NCT03706456
Title: A Phase 3, Multicenter, Open-Label, Uncontrolled Study to Evaluate the Efficacy and Safety of Cx601 in the Treatment of Complex Perianal Fistulas in Adult Patients With Crohn's Disease
Brief Title: Phase 3 Study of Cx601 in Participants With Complex Perianal Fistulising Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Darvadstrocel-3002; U1111-1218-8079 (Other: WHO); JapicCTI-184145 (Registry Identifier: JapicCTI); Alofisel-3002 (Other: Takeda)
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Results first posted 2021-10-07 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Complex Perianal Fistulas in Adult Participants With Crohn's Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Darvadstrocel 24 mL (Experimental): Darvadstrocel (Cx601) 24 mL suspension of 120 million cells of expanded allogeneic adipose-derived stem cells (eASC) as an intralesional injection, once on Day 1.
  Interventions: Biological: Darvadstrocel

INTERVENTIONS:
Biological: Darvadstrocel — Darvadstrocel cell suspension for intralesional injection.
  Other Names: Cx601

SUMMARY:
The purpose of this study is to evaluate the efficacy of darvadstrocel for the treatment of complex perianal fistulas in adult participants with Crohn's disease over 24 weeks.

DETAILED DESCRIPTION:
The drug being tested in this study is called Darvadstrocel (Cx601). This study will assess the efficacy for 24 and 52 weeks, and safety for 156 weeks of darvadstrocel when administered with intralesional injection in adult participants with Crohn's disease whose complex perianal fistulas were previously treated and refractory.

The study enrolled 22 participants. All participants who will meet the criteria will be assigned to screening period for approximately 5 weeks and after that will be enrolled the treatment period which will be the day of study product administration. After the treatment period, this study will include the follow-up period for approximately 52 weeks after study product administration, and the long-term follow-up period from Week 52 to Week 156.

This multi-center trial will be conducted in Japan. The overall time to participate is totally approximately 156 weeks (3 years) from the start of treatment period plus follow-up and long-term follow-up period. Participants will make multiple visits to the clinic and a final visit 156 weeks after treatment of study product for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with the protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. The participant who was diagnosed with Crohn's disease at least 6 months prior to the screening period according to the Diagnostic Criteria for Crohn's Disease issued by Research Group for Intractable Inflammatory Bowel Disease Designated as Specified Disease by the Ministry of Health, Labour and Welfare (MHLW) of Japan (revised January 2017).
4. The participant is either a male or female outpatient, aged 18 years or older at the time of signing the informed consent form.
5. The participant who has non-active or mildly active Crohn's disease defined by the Crohn's disease activity index (CDAI) =<220 evaluated at any time between Visit 1 and Visit 2.
6. The participant who has complex perianal fistulas with a maximum of 2 internal openings and a maximum of 3 external openings, confirmed by clinical assessment and MRI. All of the external openings must connect to internal openings. Fistula must have been draining for at least 6 weeks prior to the screening. Complex perianal fistula is defined as the one that meets 1 or more of the following criteria:

   * High (ie, above the dentate line) inter-sphincteric or trans-sphincteric fistula, extrasphincteric fistula, or supra-sphincteric fistula.
   * Presence of >=2 external openings (tracts).
   * Associated fluid collections.
7. The participant whose perianal fistulas were previously treated and have shown an inadequate response (absence of closure of part or all fistula tract, or new fistula during induction treatment) or a loss of response (fistula relapse after complete closure of initial fistula, or fistula worsening after partial closure of initial fistula during maintenance treatment) while they were receiving either immunosuppressants or biologics, or having documented intolerance (occurrence, at any time, of an unacceptable level of treatment-related side effects that makes necessary treatment discontinuation) to any of these treatments administered at least approved or recommended doses during the minimum period mentioned;

   * Antibiotics (ciprofloxacin or metronidazole): 1 or more month treatment.
   * Immunosuppressants (azathioprine, 6-mercaptopurine or methotrexate): 3 or more months treatment.
   * Biologics (anti-tumor necrosis factors [TNFs], anti-integrin or anti-interleukin [IL]-12/23): 14 or more weeks (16 or more weeks for anti-IL-12/23) standard treatment for induction or maintenance.
8. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent up to Week 52 of the study.
9. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent up to Week 52 of the study.

Exclusion Criteria:

1. The participant whose CDAI is >220 at any time between Visit 1 and Visit 2, or who has active Crohn's disease requiring a new of escalating immediate therapy.
2. The participant who has concomitant rectovaginal or rectovesical fistulas.
3. The participant who has >2 internal openings of >3 external openings.
4. The participant who is naïve to protocol required treatment for complex perianal fistulising Crohn's disease (ie, antibiotics, immunosuppressants or biologics).
5. The participant who has an abscess or collections >2 cm.
6. The participant who has rectal and/or anal stenosis and/or active proctitis, which would restrict the surgical procedure.
7. The participant who underwent surgery other than drainage or seton placement for the to be treated fistula.
8. The participant who has diverting stomas.
9. The participant who was treated with systemic steroids in the 4 weeks prior to study product administration.
10. The participant receiving cytapheresis therapy.
11. The participant who requires new treatment with immunosuppressants/biologics/non-tapered systematic steroids during the screening period.
12. The participant who has renal impairment defined by creatinine clearance below 60 mL/minute calculated using Cockcroft-Gault formula or by serum creatinine >=1.5 × upper limit of normal (ULN).
13. The participant who has hepatic impairment defined by both total bilirubin >=1.5 × ULN, and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) >=2.5 × ULN.
14. The participant who has history of abuse of alcohol or other addictive substances in the 6 months prior to the screening period.
15. The participant who has malignant tumour or who has a history of malignant tumour, including any type of fistula carcinoma.
16. The participant who has abnormal, severe, progressive, uncontrolled hepatic, hematological, gastrointestinal (except Crohn's disease), endocrine, pulmonary, cardiac, neurological, psychiatric, or cerebral disease, or the participant who developed any of the above diseases within 3 months prior to the screening period.
17. The participant who has congenital or acquired immunodeficiency, including participants known to be Human Immunodeficiency Virus (HIV) carriers.
18. The participant who has clinically significant chronically active hepatopathy of any origin, including hepatic cirrhosis, and participants who is persistent positive for hepatitis B virus (HBV) surface antigen (HBsAg) and quantitative HBV polymerase chain reaction (PCR), or positive serology for hepatitis C virus (HCV) and quantitative HCV-PCR within 6 months prior to the screening period.
19. The participant who has known allergies or hypersensitivity to antibiotics (including but not limited to penicillin, streptomycin, gentamicin, aminoglycosides), Human Serum Albumin (HSA), bovine-derived materials, local anesthetics or gadolinium (MRI contrast agent).
20. The participant for whom MRI scan is contraindicated (eg, due to the presence of a pacemaker, a history of hip replacements, or severe claustrophobia).
21. The participant who has major surgery (eg, surgery under general anesthesia, laparotomy, thoracotomy, craniotomy) or severe trauma within 6 months prior to the screening period.
22. The female participant who is pregnant, or is lactating.
23. The participant who has received any investigational drug within 12 weeks (84 days) prior to the screening.
24. The participant who has received expanded allogeneic adipose-derived stem cells (eASC) in a previous clinical study or as a therapeutic agent.
25. The participant who needs perianal surgery other than fistulas preparation required by the protocol during the screening, or the participant who will receive a perianal surgery within 24 weeks after study product administration.
26. The participant for whom anesthesia is contraindicated.
27. The participant who received excluded medications or treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2023-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (11):
- Japan (11):
  - Ieda Hospital, Toyota, Aichi-ken
  - Fukuoka University Chikushi Hospital, Chikushino-shi, Fukuoka
  - Sapporo Higashi Tokushukai Hospital, Sapporo, Hokkaido
  - Hyogo College of Medicine, Nishinomiya, Hyōgo
  - Yokohama Municipal Citizen's Hospital, Yokohama, Kanagawa
  - Mie University Hospital, Tsu, Mie-ken
  - Tohoku Rosai Hospital, Sendai, Miyagi
  - Tohoku University Hospital, Sendai, Miyagi
  - Osaka University Hospital, Suita, Osaka
  - JCHO Tokyo Yamate Medical Center, Shinjuku, Tokyo
  - Coloproctology Center Takano Hospital, Kumamoto

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Furukawa S, Mizushima T, Nakaya R, Shibata M, Yamaguchi T, Watanabe K, Futami K. Darvadstrocel for Complex Perianal Fistulas in Japanese Adults with Crohn's Disease: A Phase 3 Study. J Crohns Colitis. 2023 Apr 3;17(3):369-378. doi: 10.1093/ecco-jcc/jjac144. PMID 36149832
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b60224db2bf003ab49683

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 9 investigative sites in Japan from 06 March 2019 to 10 February 2023.
Pre-assignment Details: Participants with a diagnosis of complex perianal fistulising Crohn's disease were enrolled to receive darvadstrocel once daily.
Period: Overall Study
Arm/Group | Darvadstrocel 24 mL
Started | 22
Completed | 19
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) Population included all participants enrolled in the study.
Groups:
- Darvadstrocel 24 mL: Darvadstrocel (Cx601) 24 mL suspension of 120 million cells of eASC as an intralesional injection, once on Day 1.
Arm/Group | Darvadstrocel 24 mL
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (10.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 22
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 166.0 (8.28)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 68.33 (23.102)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — BMI=weight (kg)/[height (m)^2].
  kilogram per square meter (kg/m^2) | 24.59 (7.186)
Smoking Classification [Count of Participants; unit: Participants]
  Participants has Never Smoked | 16
  Participants is a Current Smoker | 2
  Participants is an Ex-Smoker | 4
Duration of Crohn's Disease [Mean (Standard Deviation); unit: years] — Duration of Crohn's Disease (years) is calculated by (Date of informed consent - Date of CD Diagnosis) divided by 365.25.
  years | 11.3 (6.64)
Concomitant Medications [Count of Participants; unit: Participants] — Number of participants who administered concomitant medications such as biologics, immunosuppressants, biologics plus immunosuppressants, and none of two types of concomitant drugs were reported.
  Participants
    Biologics Only | 9
    Immunosuppressants Only | 2
    Biologics+Immunosuppressants | 7
    None of 2 Types of Concomitant Drugs | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Combined Remission of Perianal Fistulising Crohn's Disease (CD) at Week 24
Description: Combined remission of perianal fistulising CD is defined as the clinically confirmed closure of all treated external openings that were draining at Screening despite gentle finger compression, and absence of collections >2 cm in the treated fistulas, confirmed by central magnetic resonance imaging (MRI) assessment at Week 24 visit. In case of missing values, last observation carried forward (LOCF) method was applied. Percentages are rounded off to the nearest decimal point.
Time Frame: Week 24
Population: ITT Population included all participants enrolled in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Darvadstrocel 24 mL
Number analyzed (Participants) | 22
percentage of participants | 59.1 [38.5 to 79.6]

2. Secondary Outcome: Percentage of Participants With Clinical Remission of Perianal Fistulising CD at Week 24
Description: Clinical remission of perianal fistulising CD is defined as the clinically confirmed closure of all treated external openings that were draining at Screening despite gentle finger compression at Week 24 Visit. In case of missing values, LOCF method was applied. Percentages are rounded off to the nearest decimal point.
Time Frame: Week 24
Population: ITT Population included all participants enrolled in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Darvadstrocel 24 mL
Number analyzed (Participants) | 22
percentage of participants | 59.1 [38.5 to 79.6]

3. Secondary Outcome: Percentage of Participants With Response of Perianal Fistulising CD at Week 24
Description: Response of perianal fistulising CD is defined as the clinically confirmed closure of at least 50 percent of all treated external openings that were draining at Screening despite gentle finger compression at Week 24 visit. In case of missing values, LOCF method was applied. Percentages are rounded off to the nearest decimal point.
Time Frame: Week 24
Population: ITT Population included all participants enrolled in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Darvadstrocel 24 mL
Number analyzed (Participants) | 22
percentage of participants | 81.8 [65.7 to 97.9]

4. Secondary Outcome: Time to Clinical Remission of Perianal Fistulising CD by Week 24
Description: Time to clinical remission is defined as the time from the study product administration to the first visit by which clinical remission is observed. Clinical remission is defined as the clinically confirmed closure of all treated external openings that were draining at Screening despite gentle finger compression.
Time Frame: Up to Week 24
Population: ITT Population included all participants enrolled in the study. Overall number of participants analyzed are the participants with clinical remission at least once during the 24-week period.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Darvadstrocel 24 mL
Number analyzed (Participants) | 16
days | 30.0 [14.0 to 116.0]

5. Secondary Outcome: Time to Response of Perianal Fistulising CD by Week 24
Description: Time to response is defined as the time from the study product administration to the first visit by which response is observed. Response is defined as the clinically confirmed closure of at least 50 percent of all treated external openings that were draining at Screening despite gentle finger compression.
Time Frame: Up to Week 24
Population: ITT Population included all participants enrolled in the study. Overall number of participants analyzed are the participants with response at least once during the 24-week period.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Darvadstrocel 24 mL
Number analyzed (Participants) | 19
days | 18.0 [12.0 to 30.0]

6. Secondary Outcome: Percentage of Participants With Relapse of Perianal Fistulising CD at Week 24 in Participants With Clinical Remission at a Previous Visit
Description: Relapse is defined as the clinically confirmed reopening of any of the treated external openings with active drainage, or the development of a collection >2 cm in the treated fistulas confirmed by central MRI assessment in participants who achieved clinical remission before Week 24. LOCF method was applied. Percentages are rounded off to the nearest decimal point.
Time Frame: Week 24
Population: ITT Population included all participants enrolled in the study. Overall number of participants analyzed are the participants who achieved clinical remission.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Darvadstrocel 24 mL
Number analyzed (Participants) | 16
percentage of participants | 25.0 [3.8 to 46.2]

7. Secondary Outcome: Time to Relapse of Perianal Fistulising CD by Week 24 in Participants With Clinical Remission at a Previous Visit
Description: Time to Relapse is defined as the time from the first visit by which clinical remission is observed to the first visit by which relapse is observed. Relapse is defined as the clinically confirmed reopening of any of the treated external openings with active drainage, or the development of a collection >2 cm in the treated fistulas confirmed by central MRI assessment.
Time Frame: Up to Week 24
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Darvadstrocel 24 mL
Number analyzed (Participants) | 16
days | NA [85.0 to NA] — Median and upper limit of 95% confidence interval was not evaluated due to insufficient number of participants with relapse.

8. Secondary Outcome: Change From Baseline in Perianal Disease Activity Index (PDAI): Total Score at Week 24
Description: The PDAI is a scoring system to evaluate the severity of perianal lesion associated with Crohn's disease. It includes the following 5 items: (a) Discharge; (b) Pain; (c) Restriction of sexual activity; (d) Type of perianal disease; and (e) Degree of induration. Each item is graded on a 5-point scale where 0 indicates no symptoms and 4 indicates severe symptoms and total range of score is from 0 to 20. Higher score indicates more severe disease. Negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 24
Population: ITT Population included all participants enrolled in the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Darvadstrocel 24 mL
Number analyzed (Participants) | 22
score on a scale
  Baseline | 4.8 (2.15)
  Change from Baseline at Week 24 | -2.4 (2.22)

9. Secondary Outcome: Change From Baseline in PDAI: Discharge Sub-Score at Week 24
Description: The PDAI is a scoring system to evaluate the severity of perianal lesion associated with Crohn's disease. It includes the following 5 items: (a) Discharge; (b) Pain; (c) Restriction of sexual activity; (d) Type of perianal disease; and (e) Degree of induration. The discharge item is graded on a 5-point scale where 0 indicates no symptoms and 4 indicates severe symptoms and total range of score is from 0 to 4. Higher score indicates more severe disease. Negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 24
Population: ITT Population included all participants enrolled in the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Darvadstrocel 24 mL
Number analyzed (Participants) | 22
score on a scale
  Baseline | 0.9 (0.64)
  Change from Baseline at Week 24 | -0.4 (0.79)

10. Secondary Outcome: Change From Baseline in PDAI: Pain Sub-Score at Week 24
Description: The PDAI is a scoring system to evaluate the severity of perianal lesion associated with Crohn's disease. It includes the following 5 items: (a) Discharge; (b) Pain; (c) Restriction of sexual activity; (d) Type of perianal disease; and (e) Degree of induration. The pain item is graded on a 5-point scale where 0 indicates no symptoms and 4 indicates severe symptoms and total range of score is from 0 to 4. Higher score indicates more severe disease. Negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 24
Population: ITT Population included all participants enrolled in the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Darvadstrocel 24 mL
Number analyzed (Participants) | 22
score on a scale
  Baseline | 0.9 (0.92)
  Change from Baseline at Week 24 | -0.6 (0.90)

11. Secondary Outcome: Change From Baseline in Crohn's Disease Activity Index (CDAI): Total Score at Week 24
Description: CDAI score is calculated from the following 8 items: (a) Number of liquid or very soft stools; (b) Abdominal pain; (c) General wellbeing; (d) Extraintestinal complications; (e) Antidiarrhoeal drugs; (f) Abdominal mass; (g) Hematocrit; and (h) Body weight. Scores of some items in CDAI are calculated based on patient diary. Total score ranges from 0 to 600. Higher score means more severe disease and especially severe disease was defined as a value of greater than 450. Negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 24
Population: ITT Population included all participants enrolled in the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Darvadstrocel 24 mL
Number analyzed (Participants) | 22
score on a scale
  Baseline | 94.25 (60.048)
  Change from Baseline at Week 24 | -5.15 (47.500)

12. Secondary Outcome: Change From Baseline in Van Assche Score at Week 24
Description: The Van Assche score represents the magnetic resonance imaging (MRI)- based severity of perianal lesion associated with Crohn's disease. Based on MRI data, the number, location and extension of fistula tracts, hyperintensity on T2-weighted images, presence or absence of collections (cavities >3 mm in diameter), and rectal wall involvement will be evaluated. The score range was from 0 to 22. Higher score means more severe disease. Negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 24
Population: ITT Population included all participants enrolled in the study. Overall number of participants analyzed were participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Darvadstrocel 24 mL
Number analyzed (Participants) | 18
score on a scale
  Baseline | 14.5 (3.99)
  Change from Baseline at Week 24 | -1.7 (4.35)

13. Secondary Outcome: Percentage of Participants With Combined Remission of Perianal Fistulising CD at Week 52
Description: Combined remission is defined as the clinically confirmed closure of all treated external openings that were draining at the screening despite gentle finger compression, and absence of collections >2 cm in the treated fistulas which is confirmed by the central MRI assessment at Week 52 visit. In case of missing values, LOCF method was applied. Percentages are rounded off to the nearest decimal point.
Time Frame: Week 52
Population: ITT Population included all participants enrolled in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Darvadstrocel 24 mL
Number analyzed (Participants) | 22
percentage of participants | 68.2 [48.7 to 87.6]

14. Secondary Outcome: Percentage of Participants With Clinical Remission of Perianal Fistulising CD at Week 52
Description: Clinical remission is defined as the clinically confirmed closure of all treated external openings that were draining at screening despite gentle finger compression at Week 52 visit. In case of missing values, LOCF method was applied. Percentages are rounded off to the nearest decimal point.
Time Frame: Week 52
Population: ITT Population included all participants enrolled in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Darvadstrocel 24 mL
Number analyzed (Participants) | 22
percentage of participants | 72.7 [54.1 to 91.3]

15. Secondary Outcome: Percentage of Participants With Response of Perianal Fistulising CD at Week 52
Description: Response is defined as the clinically confirmed closure of at least 50 percent of all treated external openings that were draining at the screening despite gentle finger compression at Week 52 visit. In case of missing values, LOCF method was applied. Percentages are rounded off to the nearest decimal point.
Time Frame: Week 52
Population: ITT Population included all participants enrolled in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Darvadstrocel 24 mL
Number analyzed (Participants) | 22
percentage of participants | 90.9 [78.9 to 100.0]

16. Secondary Outcome: Time to Combined Remission of Perianal Fistulising CD by Week 52
Description: Time to combined remission is defined as the time from the study product administration to the first visit by which combined remission is observed. Combined remission is defined as the clinically confirmed closure of all treated external openings that were draining at the screening despite gentle finger compression, and absence of collections >2 cm in the treated fistulas which is confirmed by the central MRI assessment.
Time Frame: Up to Week 52
Population: ITT Population included all participants enrolled in the study. Overall number analyzed is the number of participants who achieved combined remission at least once during the 52-week period.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Darvadstrocel 24 mL
Number analyzed (Participants) | 17
days | 175.5 [165.0 to 365.0]

17. Secondary Outcome: Time to Clinical Remission of Perianal Fistulising CD by Week 52
Description: as for outcome 4
Time Frame: Up to Week 52
Population: ITT Population included all participants enrolled in the study. Overall number analyzed is the number of participants who achieved clinical remission at least once during the 52-week period.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Darvadstrocel 24 mL
Number analyzed (Participants) | 20
days | 25.5 [14.0 to 109.0]

18. Secondary Outcome: Time to Response of Perianal Fistulising CD by Week 52
Description: Time to response is defined as the time from the study product administration to the first visit by which response is observed. Response is defined as the clinically confirmed closure of at least 50 percent of all treated external openings that were draining at the Screening despite gentle finger compression.
Time Frame: Up to Week 52
Population: ITT Population included all participants enrolled in the study. Overall number analyzed is the number of participants who achieved response at least once during the 52-week period.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Darvadstrocel 24 mL
Number analyzed (Participants) | 21
days | 18.0 [12.0 to 30.0]

19. Secondary Outcome: Percentage of Participants With Relapse of Perianal Fistulising CD at Week 52 in Participants With Combined Remission at Week 24
Description: Relapse is defined as the clinically confirmed reopening of any of the treated external openings with active drainage, or the development of a collection >2 cm in the treated fistulas confirmed by central MRI assessment in participants who achieved combined remission at Week 24. Combined remission is defined as the clinically confirmed closure of all treated external openings that were draining at Screening despite gentle finger compression, and absence of collections >2 cm in the treated fistulas, confirmed by the central MRI assessment. LOCF method was applied. Percentages are rounded off to the nearest decimal point.
Time Frame: Week 52
Population: ITT Population included all participants enrolled in the study. Overall number analyzed is the number of participants with combined remission at Week 24.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Darvadstrocel 24 mL
Number analyzed (Participants) | 13
percentage of participants | 23.1 [0.2 to 46.0]

20. Secondary Outcome: Time to Relapse of Perianal Fistulising CD by Week 52 in Participants With Combined Remission at Week 24
Description: Time to relapse by Week 52 in participants who achieved combined remission at Week 24 is defined as the time from the combined remission at Week 24 to the first visit by which relapse is observed. Relapse is defined as the clinically confirmed reopening of any of the treated external openings with active drainage, or the development of a collection >2 cm in the treated fistulas confirmed by central MRI assessment in participants who achieved combined remission at Week 24. Combined remission is defined as the clinically confirmed closure of all treated external openings that were draining at Screening despite gentle finger compression, and absence of collections >2 cm in the treated fistulas, confirmed by the central MRI assessment.
Time Frame: Up to Week 52
Population: as for outcome 19
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Darvadstrocel 24 mL
Number analyzed (Participants) | 13
days | NA [NA to NA] — Median, lower and upper limits of confidence interval was not estimable due to low number of participants with relapse..

21. Secondary Outcome: Change From Baseline in PDAI: Total Score at Week 52
Description: The PDAI is a scoring system to evaluate the severity of perianal lesion associated with Crohn's disease. It includes the following 5 items: (a) Discharge; (b) Pain; (c) Restriction of sexual activity; (d) Type of perianal disease; and (e) Degree of induration. Each item is graded on a 5-point scale ranging from no symptoms (score of 0) to severe symptoms (score of 4) and total range of score is from 0 to 20. Higher score indicates more severe disease. Negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 52
Population: ITT Population included all participants enrolled in the study. Overall number analyzed is the number of participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Darvadstrocel 24 mL
Number analyzed (Participants) | 20
score on a scale | -2.8 (2.59)

22. Secondary Outcome: Change From Baseline in PDAI: Discharge Sub-Score at Week 52
Description: The PDAI is a scoring system to evaluate the severity of perianal lesion associated with Crohn's disease. It includes the following 5 items: (a) Discharge; (b) Pain; (c) Restriction of sexual activity; (d) Type of perianal disease; and (e) Degree of induration. The discharge item is graded on a 5-point scale ranging from no symptoms (score of 0) to severe symptoms (score of 4) and total range of score is from 0 to 20. Higher score indicates more severe disease. Negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Darvadstrocel 24 mL
Number analyzed (Participants) | 20
score on a scale | -0.5 (0.95)

23. Secondary Outcome: Change From Baseline in PDAI: Pain Sub-Score at Week 52
Description: The PDAI is a scoring system to evaluate the severity of perianal lesion associated with Crohn's disease. It includes the following 5 items: (a) Discharge; (b) Pain; (c) Restriction of sexual activity; (d) Type of perianal disease; and (e) Degree of induration. The pain item is graded on a 5-point scale ranging from no symptoms (score of 0) to severe symptoms (score of 4) and total range of score is from 0 to 20. Higher score indicates more severe disease. Negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Darvadstrocel 24 mL
Number analyzed (Participants) | 20
score on a scale | -0.8 (1.06)

24. Secondary Outcome: Change From Baseline in CDAI: Total Score at Week 52
Description: CDAI score is calculated from the following 8 items: (a) Number of liquid or very soft stools; (b) Abdominal pain; (c) General wellbeing; (d) Extraintestinal complications; (e) Antidiarrhoeal drugs; (f) Abdominal mass; (g) Hematocrit; and (h) Body weight. Scores of some items in CDAI are calculated based on patient diary. Total score ranges from 0 to 600. Higher score indicates more severe disease and especially severe disease was defined as a value of greater than 450. Negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Darvadstrocel 24 mL
Number analyzed (Participants) | 21
score on a scale | -20.86 (51.331)

25. Secondary Outcome: Change From Baseline in Van Assche Total Score at Week 52
Description: The Van Assche score represents the MRI-based severity of perianal lesion associated with Crohn's disease. Based on MRI data, the number, location and extension of fistula tracts, hyperintensity on T2-weighted images, presence or absence of collections (cavities >3 mm in diameter), and rectal wall involvement will be evaluated. The total score ranges from 0 to 22. Higher score indicates more severe disease. Negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Darvadstrocel 24 mL
Number analyzed (Participants) | 17
score on a scale | -2.2 (4.90)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Week 156
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Darvadstrocel 24 mL
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 11/22
Other Adverse Events (participants affected / at risk) | 18/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Darvadstrocel 24 mL (N=22)
Anal fistula (Gastrointestinal disorders) | 1
COVID-19 (Infections and infestations) | 4
Calculus urinary (Renal and urinary disorders) | 1
Crohn's disease (Gastrointestinal disorders) | 3
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Premature labour (Pregnancy, puerperium and perinatal conditions) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Darvadstrocel 24 mL (N=22)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Anal fistula (Gastrointestinal disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 3
Cheilitis (Gastrointestinal disorders) | 2
Dental caries (Gastrointestinal disorders) | 2
Fistula (Musculoskeletal and connective tissue disorders) | 2
Nasopharyngitis (Infections and infestations) | 6
Nausea (Gastrointestinal disorders) | 2
Pharyngitis (Infections and infestations) | 2
Proctalgia (Gastrointestinal disorders) | 7
Pyrexia (General disorders) | 2
Rhinitis (Infections and infestations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/56/NCT03706456/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT03706456/SAP_002.pdf